CLINICAL TRIAL: NCT06190171
Title: Impact of Preoperative Respiratory Strength Training on Postoperative Health for Heart Transplant Recipients
Brief Title: Respiratory Strength Training in Heart Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cara Donohue, Ph.D. CCC-SLP, Assistant Professor, Director of Medical Speech-Language Pathology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 232071; 24CDA1257668 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2023-12-01; First posted 2024-01-05 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Dysphagia; Heart Transplant Recipients
Keywords: dysphagia; deglutition; deglutition disorders; swallowing; breathing; cough; swallowing disorders; heart transplant recipients; respiratory muscle strength training
MeSH Terms: conditions — Deglutition Disorders; Respiratory Aspiration; Cough

STUDY DESIGN:
Intervention Model Description: randomized, sham controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be assigned to active or sham respiratory strength training using block randomization and will be blinded to their assigned treatment. Researchers performing evaluations and data analysis will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active respiratory muscle strength training (Experimental): Enrolled heart transplant patients will undergo active preoperative respiratory strength training using two respiratory strength training devices from enrollment until they receive a heart transplant.
  Interventions: Behavioral: Active respiratory muscle strength training
- Sham respiratory muscle strength training (Sham Comparator): Enrolled heart transplant patients will undergo sham preoperative respiratory strength training using two respiratory strength training devices from enrollment until they receive a heart transplant. For individuals completing sham respiratory strength training, the spring will be removed from the devices as has been done in prior sham-controlled trials.
  Interventions: Behavioral: Sham respiratory muscle strength training

INTERVENTIONS:
Behavioral: Active respiratory muscle strength training — Devices will be set to 60% of participants' maximum expiratory pressure and maximum inspiratory pressure. Participants will complete training 7 days per week by performing 5 sets of 5 repetitions for both expiratory and inspiratory muscle strength training (a total of 50 repetitions).
  Arms: Active respiratory muscle strength training
Behavioral: Sham respiratory muscle strength training — Springs will be removed from devices to ensure training is done without resistance. Participants will complete training 7 days per week by performing 5 sets of 5 repetitions for both expiratory and inspiratory sham muscle strength training (a total of 50 repetitions).
  Arms: Sham respiratory muscle strength training

SUMMARY:
This research study is investigating whether completing breathing exercises before surgery helps heart transplant patients recover after surgery. Previous studies have shown that breathing exercises can improve breathing, cough, and swallow function in patients with other diseases/conditions. The current study will investigate the impact of a preoperative respiratory muscle strength training program on breathing and cough function, swallow function, patient-reported eating and swallowing fatigue, and health outcomes in individuals undergoing heart transplantation.

Participants will:

* undergo tests of breathing, cough, and swallow function
* complete questionnaires about the treatment, their swallow function
* complete breathing exercises daily

DETAILED DESCRIPTION:
This study will involve three in-person research evaluations to our lab or in the hospital that will last 45 minutes- 1 hour and will consist of a screening, breathing and cough testing, swallow function testing, and completion of questionnaires. Following the initial research evaluation, individuals will complete daily exercises of active or sham respiratory muscle strength training for several weeks with one telehealth or in-person session per week. The exercises will take 10-15 minutes to complete, and individuals will fill out training logs daily. Prior to transplantation and after completion of the breathing exercises, individuals will undergo a second research evaluation. Then, following surgery, individuals will undergo a third research evaluation and outcomes will be tracked via the electronic health records system.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (18-90 years old)
2. Not pregnant
3. Undergoing evaluation or actively waitlisted for heart transplantation at VUMC with a waitlist status of 1-6
4. Have a computer, tablet or electronic device with a stable internet connection for telehealth sessions (outpatient)
5. Be willing to undergo testing procedures and complete the exercise training program.

Exclusion Criteria:

1. Individual <18 years old, >90 years old
2. Pregnant
3. No access to a computer, tablet or electronic device with a stable internet connection for telehealth sessions
4. Unwilling or unable to undergo testing procedures and complete the exercise training program.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in maximum expiratory pressure between pre and post respiratory strength training | baseline, post-intervention/pre-surgery (an average of 2-6 weeks after baseline)
  A measure of respiratory strength while breathing out
Change in maximum inspiratory pressure between pre and post respiratory strength training | baseline, post-intervention/pre-surgery (an average of 2-6 weeks after baseline)
  A measure of respiratory strength while breathing in

SECONDARY OUTCOMES:
Change in cough peak expiratory flow between pre and post respiratory strength training | baseline, post-intervention/pre-surgery (an average of 2-6 weeks after baseline)
  A measure of cough strength
Patient-reported treatment burden | post-intervention/pre-surgery (an average of 2-6 weeks after baseline)
  Patients will complete the exercise therapy burden questionnaire (ETBQ). Scores on the ETBQ range from 0-100 with higher scores indicating greater burden.
Patient reported swallow function | pre-surgery (baseline), post-surgery
  Patients will complete the swallowing and eating related fatigue (SERF) questionnaire. Scores on the SERF range from 0-48 with higher scores indicating greater impairment.
Change in penetration-aspiration scale scores between before and after surgery | pre-surgery (baseline), post-surgery
  The penetration aspiration scale is a validated 8-point ordinal rating scale that measures the depth of airway invasion and the patient's response during swallowing. Scores range from 1 to 8 with a score of 1 indicating a safe swallow (best score) and 8 indicating silent aspiration (worst score).
Change in clinical frailty scale score | baseline, post-intervention/pre-surgery (an average of 2-6 weeks after baseline)
  The Clinical Frailty Scale (CFS) is a measure of physical function. Scores on the CFS range from 1-9 with higher scores indicating greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Donohue, Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT06190171/ICF_001.pdf